CLINICAL TRIAL: NCT00720395
Title: Predictors of Postpartum Relapse in Women With Bipolar Disorder
Brief Title: Identifying Predictors of Bipolar Disorder Relapse During Pregnancy and the Postpartum Period
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn [Funding was never granted for this study. No participants were ever enrolled.]
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Donald Jeffery Newport, MD, Emory University
Other Study IDs: R01 MH085026; DATR A2-AIE
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2009-03

CONDITIONS: Bipolar Disorder
Keywords: Psychiatry; Pregnancy
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, and urine samples are processed and stored at each study visit.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Women with bipolar disorder who are preconception or pregnant. Primary focus on predictors of postpartum bipolar disorder relapse and burden of illness through first six months postpartum

SUMMARY:
This study will evaluate pregnant women who have bipolar disorder to gain a better understanding of risk factors for bipolar disorder relapse during pregnancy and the postpartum period.

DETAILED DESCRIPTION:
Bipolar disorder, also known as manic-depressive illness, is a brain disorder that causes significant changes in a person's mood and energy. The onset of bipolar disorder usually occurs during young adulthood and persists for the rest of a person's life, making women who are of childbearing age at risk for this disorder. Although overall relapse rates for pre-existing mood disorders are typically higher in women who are pregnant or recently gave birth than in other women, very little is known about the impact of pregnancy and the postpartum period on someone with bipolar disorder. The course and treatment of maternal mental illness during pregnancy and the postpartum period remains the center of much debate, particularly with respect to the use of psychotropic medications during pregnancy and breastfeeding. Identifying predictors of bipolar disorder recurrence during pregnancy and the postpartum period may help to determine which women are at highest risk and to develop new treatment guidelines. However, more information is needed to both identify predictors and develop guidelines that will improve outcomes for pregnant women with bipolar disorder and their babies. This study will evaluate pregnant women who have bipolar disorder to gain a better understanding of risk factors for bipolar disorder relapse during pregnancy and the postpartum period.

Participation in this study will last up to 6 months postpartum. Study visits will be scheduled every 4 weeks during pregnancy and every 6 weeks after delivery for up to 6 months postpartum. During study visits, data will be collected on factors that may predict bipolar disorder recurrence and overall burden of bipolar disorder illness. Specific potential factors that will be evaluated include severity of illness in the past, type and severity of both recent and past life stressors, and any treatment received during pregnancy and the postpartum period. The study will also evaluate how antidepressant medications, if taken, affect the mother and baby during pregnancy and the postpartum period. Additionally, plasma, serum, and urine samples will also be processed and stored at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* Meets DSM-IV criteria for bipolar disorder of any subtype
* No more than 32 weeks gestation, dated by last menstrual period

Exclusion Criteria:

* Active suicidality or homicidality
* Acute psychotic symptoms

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include women who are pregnant or recently gave birth and who meet DSM-IV criteria for any subtype of bipolar disorder.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Preconception, predelivery, and postpartum predictors of postpartum bipolar disorder relapse and burden of illness | Measured at Year 1 postpartum

SECONDARY OUTCOMES:
Impact of predelivery expectations, the role of breastfeeding, and self-reported sleep disturbance in the risk for postpartum bipolar disorder relapse | Measured at Year 1 postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Donald J. Newport, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Psychaitry and Behavioral Sciences, Atlanta, Georgia, United States

REFERENCES:
- See also: Click here for more information on this study at Emory University's Women's Mental Health Program site — http://emorywomensprogram.org